CLINICAL TRIAL: NCT03675932
Title: Rapid Cadence Cycling for Parkinson's Disease: A Study of Implementation and Efficacy in the Community Setting
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: The Cleveland Clinic (Other)
Responsible Party: Principal Investigator, Anne-Marie Alexandra Wills, MD, Assistant Professor in Neurology, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2018P001116
Record Dates: First submitted 2018-09-08; First posted 2018-09-18 (Actual); Last update posted 2020-02-25 (Actual); Status verified 2020-02

CONDITIONS: Parkinson Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Cycling Intervention (Experimental): Single-arm trial. All participants will receive the same intervention of Rapid Cadence Cycling on a Solo-Rider Spin Bicycle
  Interventions: Other: Rapid Cadence Cycling on a Solo-Rider Spin Bicycle

INTERVENTIONS:
Other: Rapid Cadence Cycling on a Solo-Rider Spin Bicycle — Individuals with Parkinson's Disease will participate in 60 minute spin-classes during which they will follow the Pedaling for Parkinson's(TM) Foundation recommended protocol to achieve a cadence of 80-90 during the 40 minute main set.

SUMMARY:
Forced cadence cycling (FCC) in which individuals with Parkinson's Disease (PD) pedal with external augmentation at 80-90 revolutions per minute (rpm) has demonstrated significant motor improvement in prior clinical trials. These studies required either a tandem bicycle with second rider or an expensive motorized bicycle, making this therapy inaccessible to most patients. In this pragmatic open-label before and after pilot study investigators examine implementation and effectiveness of (RCC) without tandem or motor augmentation and in a community-based setting. Approximately 30 participants will be recruited to participate in 24 one-hour rapid-cadence spin classes in YMCAs over 8 weeks. Primary outcomes will examine implementation of the intervention and secondary outcomes will examine effectiveness against a historical comparison group.

ELIGIBILITY:
Inclusion Criteria:

1. Adults age 18 or older.
2. Clinically confirmed diagnosis of idiopathic PD by a movement disorder specialist.
3. Hoehn and Yahr stage I-III while ON anti-parkinsonian medication.
4. Stable or absent MAO-B inhibitors (Selegiline, Rasagiline, Zydis selegiline HCL Oral disintegrating) for at least 60 days prior to enrollment; stable or absent other medications for PD motor symptoms (Levodopa, Dopamine agonists, Anticholinergics, Amantadine, COMT-Inhibitors) for at least 30 days prior to enrollment; stable or absent medications for the following PD-non-motor symptoms: depression, anxiety, cognition, sleep, orthostatic hypotension.
5. Agreement to defer any medication changes until after completion of 8-week program and post-test measurements.
6. Written permission by a physician to participate in the program.
7. English language proficiency sufficient to understand and participate in a cycling class taught in English.

Exclusion Criteria:

1. Clinically significant medical disease that would increase the risk of exercise-related complications (eg: cardiac or pulmonary disease, uncontrolled diabetes mellitus, uncontrolled hypertension or stroke) as determined by a treating physician through letter obtained by YMCA or the study investigator.
2. Dementia as evidenced by a score of less than 116 on the Mattis Dementia Rating Scale or dementia in the opinion of the study investigator that would prohibit subject from complying with all study activities.
3. Other medical or musculoskeletal contraindication to exercise.
4. Concurrent participation in another trial of exercise therapy for PD or initiation of a new structured exercise plan during the duration of the study. Note: participants may continue any pre-existing exercise routine (including group-based classes) during the study but will be asked not to start anything new.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2018-10-01 (Actual); Primary Completion 2019-05-01 (Actual); Study Completion 2019-08-01 (Actual)

PRIMARY OUTCOMES:
Percentage of individuals who complete at least 80% of offered cycling sessions [Tolerability] | assessed at conclusion of the 8 week intervention
  Investigators will consider those who do not withdraw from the study, are not lost to follow up, and complete at least 80% of the cycling sessions to demonstrate tolerability of the study.
Proportion of subjects reporting an adverse event during class [Safety] | assessed at each class by study staff and weekly by PI for duration of 8 week intervention
  Safety will be reported descriptively and include the proportion of subjects reporting any adverse event.

SECONDARY OUTCOMES:
Modified Unified Parkinson's Disease Rating Scale-section III Motor | Assessed within two weeks prior to start of intervention and within one week after completion of intervention
  The Unified Parkinson's Disease Rating Scale (UPDRS) section III measures severity of motor symptoms of Parkinson's disease with scores ranging from 0 to 199 with higher scores indicating more severe motor symptoms. This study utilizes a modified version of the UPDRS without rigidity which will be recorded on video and rated remotely by a movement disorder neurologist blinded to intervention status of the participant. This modified version has been shown to be reliable and valid, both at cross-sectional time points and longitudinally (Abdolahi, 2013).
Timed Up and Go | Assessed within two weeks prior to start of intervention and within one week after completion of intervention
  The Timed Up and Go test is measured in seconds with a range of 5-25 seconds (longer is worse)
Trail Making Test A& B | Assessed within two weeks prior to start of intervention and within one week after completion of intervention
  This cognitive test is measured in seconds with a range (part B) of 60-240 seconds (longer is worse).
PROMIS sf v1.0 Global Health | Assessed within two weeks prior to start of intervention and within one week after completion of intervention
  A 10-item patient reported outcomes scale measuring five domains (physical function, fatigue, pain, emotional distress, social health) and general health perceptions that cut across domains. Scores can range from 0-100 where higher is better.
Assessment of Intelligibility of Dysarthria (AIDS) | Assessed within two weeks prior to start of intervention and within one week after completion of intervention
  The Assessment of Intelligibility of Dysarthric Speech is a tool for quantifying single-word intelligibility, sentence intelligibility, and speaking rate. The outcome is measured as the percent of words that are intelligible, with higher scores being better.

CONTACTS AND LOCATIONS:
Overall Officials: Anne-Marie Wills, MD, MPH, Principal Investigator — Massachusetts General Hospital; Kathleen E McKee, MD, Study Director — Massacusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No